CLINICAL TRIAL: NCT04406207
Title: Human Endogenous Retroviruses in Acute Myeloid Leukemia: Expression and Immune Impact
Brief Title: Endogenous Retroviruses in Acute Myeloid Leukemia
Acronym: ERVAL
Status: Withdrawn | Type: Observational
Why Stopped: COVID-19
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0851
Record Dates: First submitted 2020-05-13; First posted 2020-05-28 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Leukemia, Myeloid
MeSH Terms: conditions — Leukemia, Myeloid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients relapsing or not after hematopoietic stem cell transplantation.
  Interventions: Other: Demonstration of T cell responses

INTERVENTIONS:
Other: Demonstration of T cell responses — Evaluation of HERVs-specific CD8+ T cells before and after hematopoietic stem cell transplantation. Comparison will be made in patients relapsing vs non relapsing patients.
  The measurement of these responses will be done by dextramer, allowing precise and specific measurement of the lymphocytes directed against the HERVs of interest.

SUMMARY:
Allogeneic hematopoietic stem cell transplantation (HSCT) is the only curative therapy for numerous malignant hematologic diseases. Despite recent advances in the field, relapse rates are still high and the first cause of death. The identification of new relevant therapeutic targets is therefore urgently needed.

Human endogenous retroviruses (HERVs) are accounting for 8% of the human genome. While silenced at the steady state (mainly by methylation mechanisms), HERVs reactivations have been described in different conditions such as auto-immune diseases or cancer, leading to an innate and adaptive immune response. Several questions are raised in the field of hematology where few data are available, and the exact role of HERVs in these diseases is still to define.

Our team is currently working on the role of HERVs in different types of cancer. We developed a bioinformatics approach to identify overexpressed HERVs from RNAseq data. We also developed in vitro assays to assess the immunogenicity of different peptides from HERVs open reading frames and showed that several epitopes shared among different HERVs can induce a specific CD8+ T cell response. More recently, we have analyzed 151 acute myeloid leukemia (AML) RNAseq data from TCGA and identified multiple overexpressed HERVs in this disease. Immunogenicity test are currently ongoing with patient's blood at diagnosis.

The main objective of this part of our project is to analyze the establishment of a HERVs-specific CD8+ T cell response participating in graft-versus-leukemia effect after HSCT for AML patients. Secondary objectives are to analyze relations between this response and different clinical factors such as the onset of GVHD or relapse.

Peripheral blood mononuclear cells (PBMCs) from AML patients will be extracted and frozen at different time point: diagnosis, complete remission (pre-HSCT) and after HSCT (M3, M6 and M12). This prospective protocol is currently ongoing at the Centre Hospitalier Lyon Sud, with around 30 samples already available.

After having selected relevant HERVs, specific dextramers identified by DNA barcode will be synthesized. These dextramers allowing the identification of specific T cell responses directed against up to 1000 epitopes, we will be able to screen specific T cells directed against HERVs overexpressed in AML for most common HLA. Dextramer staining will be performed on PBMCs after thawing. Positive cells will be sorted by flow cytometry and DNA will be expanded by PCR before performing sequencing, allowing the identification of specific sequences by its unique DNA barcode.

The analyze of HERVs-specific CD8+ T cell responses after HSCT will allow us to better define HERVs role in the onset of graft-versus-leukemia effect. A specific T cell response without GvHD will define the relevance of such peptides as tumor specific antigens.

ELIGIBILITY:
Inclusion Criteria:

* Acute myeloid leukemia (all subtypes)
* Stem cell transplantation indication
* Non opposition to the study

Exclusion Criteria:

- Intensive care unit at diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults >= 18 years old with acute myeloid leukemia
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-01-06 (Actual); Study Completion 2022-01-06 (Actual)

PRIMARY OUTCOMES:
HERVs-specific CD8+ T cells responses | Day 0
  HERVs-specific CD8+ T cells responses will be monitored using DNA-barcode dextramers.
HERVs-specific CD8+ T cells responses | At remission <- Day 0 + 1 month
  HERVs-specific CD8+ T cells responses will be monitored using DNA-barcode dextramers.
HERVs-specific CD8+ T cells responses | Before transplant <- Day 0 + 3 month
  HERVs-specific CD8+ T cells responses will be monitored using DNA-barcode dextramers.
HERVs-specific CD8+ T cells responses | 1 month
  HERVs-specific CD8+ T cells responses will be monitored using DNA-barcode dextramers.
HERVs-specific CD8+ T cells responses | 3 months
  HERVs-specific CD8+ T cells responses will be monitored using DNA-barcode dextramers.
HERVs-specific CD8+ T cells responses | 6 months
  HERVs-specific CD8+ T cells responses will be monitored using DNA-barcode dextramers.
HERVs-specific CD8+ T cells responses | 12 months
  HERVs-specific CD8+ T cells responses will be monitored using DNA-barcode dextramers.
HERVs-specific CD8+ T cells responses | At relapse: up to 6 month after day 0
  HERVs-specific CD8+ T cells responses will be monitored using DNA-barcode dextramers.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent ALCAZER, MD, Principal Investigator — Hospices Civils de Lyon